CLINICAL TRIAL: NCT00326807
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Naltrexone in the Treatment of Concurrent Alcohol Dependence and Pathological Gambling
Brief Title: Naltrexone in the Treatment of Concurrent Alcohol Dependence and Pathological Gambling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 095/2001
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2006-05-17 (Estimated); Status verified 2006-05

CONDITIONS: Concurrent Alcohol Dependence and Pathological Gambling
Keywords: naltrexone; alcohol; gambling; concurrent
MeSH Terms: conditions — Gambling | interventions — Naltrexone

INTERVENTIONS:
Drug: Naltrexone

SUMMARY:
This study assessed whether naltrexone, an opioid antagonist, might be effective in reducing excessive gambling behavior in people who also drink heavily. The efficacy of naltrexone was evaluated in a randomized, double-blind, placebo-controlled trial. Fifty-two subjects who had significant problems with both gambling and alcohol received 11 weeks of either naltrexone or placebo.

DETAILED DESCRIPTION:
With the growing popularity of gambling, there has been an increase in the number of individuals with problem gambling. As we learn more about the way we can help problem gamblers, there is a great interest developing effective medications for this problem. Although there is much to learn about the factors that lead to gambling problems, there is some research showing that one of the reasons why gambling may be so rewarding and difficult to stop is due to the release of endogenous opioids, a specific brain chemical that is associated with the feeling of pleasure. It is possible that medications known to affect the opioidergic neurotransmitter system which produces endogenous opioids may be beneficial in reducing pathological gambling. One such medication is naltrexone, an opioid antagonist, that has been shown to be effective in reducing alcohol consumption and approved for use in the treatment of alcohol dependence. This study assessed whether naltrexone might be effective in reducing excessive gambling behavior in people who also drink heavily. The efficacy of naltrexone was evaluated in a randomized, double-blind, placebo-controlled trial. Fifty-two subjects who had significant problems with both gambling and alcohol received 11 weeks of either naltrexone or placebo. Everyone also received 7 weeks of cognitive-behavioral counselling to help them reduce or stop drinking and gambling. Changes in alcohol and gambling behavior were measured at the beginning of treatment, at the end-of-treatment and 3, 6 and 12-months after treatment follow-up. The results showed that there were no significant differences between those who received placebo versus those who received naltrexone on any alcohol or gambling measure (i.e., frequency of drinking/ gambling, amount of drinking/ gambling, money spent of gambling, urges to drink/ gamble). However, treatment in general was effective as everyone, regardless of the treatment they received, were gambling and drinking significantly less at the end-of-treatment and during the year follow-up. The conclusion of the study was that naltrexone was not an effective treatment for concurrent alcohol use and gambling problems.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of alcohol abuse and dependence
* Diagnosis of pathological gambling
* Drinking on at least 50% of the days in the preceding month
* Gambling at least weekly in the month prior to assessment

Exclusion Criteria:

* Dependence or abuse of any other psychoactive substances (except for nicotine dependence)
* Concurrent diagnoses of any other psychiatric disorder,
* Serious medical illness
* Laboratory evidence of significant hepatocellular injury
* Use of disulfiramuse and/or opioid-containing medications
* Psychosocial crisis
* Pregnancy
* Inability to read or write English.
* Poor motivation to change alcohol or gambling behavior

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2001-06; Study Completion 2004-06

PRIMARY OUTCOMES:
Gambling Urge Questionnaire
Obsessive Compulsive Drinking Scale
Readiness to Change Questionnaire
Frequency of drinking/gambling
Amount of drinking/gambling
Money spent of gambling

CONTACTS AND LOCATIONS:
Overall Officials: Tony Toneatto, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada
- National Public Health Institute, Helsinki, Finland

REFERENCES:
- [Background] Anton RF, Moak DH, Latham P, Waid LR, Myrick H, Voronin K, Thevos A, Wang W, Woolson R. Naltrexone combined with either cognitive behavioral or motivational enhancement therapy for alcohol dependence. J Clin Psychopharmacol. 2005 Aug;25(4):349-57. doi: 10.1097/01.jcp.0000172071.81258.04. PMID 16012278
- [Background] Chick J, Anton R, Checinski K, Croop R, Drummond DC, Farmer R, Labriola D, Marshall J, Moncrieff J, Morgan MY, Peters T, Ritson B. A multicentre, randomized, double-blind, placebo-controlled trial of naltrexone in the treatment of alcohol dependence or abuse. Alcohol Alcohol. 2000 Nov-Dec;35(6):587-93. doi: 10.1093/alcalc/35.6.587. PMID 11093966
- [Background] Crockford DN, el-Guebaly N. Naltrexone in the treatment of pathological gambling and alcohol dependence. Can J Psychiatry. 1998 Feb;43(1):86. No abstract available. PMID 9494755
- [Background] Feigelman W, Wallisch LS, Lesieur HR. Problem gamblers, problem substance users, and dual-problem individuals: an epidemiological study. Am J Public Health. 1998 Mar;88(3):467-70. doi: 10.2105/ajph.88.3.467. PMID 9518986
- [Background] Gianoulakis C. Endogenous opioids and excessive alcohol consumption. J Psychiatry Neurosci. 1993 Jul;18(4):148-56. PMID 7690585
- [Background] Heinala P, Alho H, Kiianmaa K, Lonnqvist J, Kuoppasalmi K, Sinclair JD. Targeted use of naltrexone without prior detoxification in the treatment of alcohol dependence: a factorial double-blind, placebo-controlled trial. J Clin Psychopharmacol. 2001 Jun;21(3):287-92. doi: 10.1097/00004714-200106000-00006. PMID 11386491
- [Derived] Dowling N, Merkouris S, Lubman D, Thomas S, Bowden-Jones H, Cowlishaw S. Pharmacological interventions for the treatment of disordered and problem gambling. Cochrane Database Syst Rev. 2022 Sep 22;9(9):CD008936. doi: 10.1002/14651858.CD008936.pub2. PMID 36130734
- See also: institution link — http://camh.net